CLINICAL TRIAL: NCT05018312
Title: Social Phobia and Evasiveness: A Feasibility, Superiority, Randomized Clinical Trial of the Effect of Modified Collaborative Assessment VS Standard Assessment on Patient's Readiness For Psychotherapy (CO-ASSM-RCT)
Brief Title: Modified Collaborative Assessment VS Standard Assessment on Readiness For Psychotherapy Among Patients With Anxiety
Acronym: CO-ASSM-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Collaborators: Research Unit for Psychotherapy and Psychopathology, Psychiatry West, Region Zealand Mental Health Service (Unknown)
Responsible Party: Principal Investigator, Sidse Arnfred, Professor, senior consultant, MD MSc PHD DMSC, Psychiatric Research Unit, Region Zealand, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021001
Record Dates: First submitted 2021-07-29; First posted 2021-08-24 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Psychotherapy; Social Anxiety Disorder; Personality Disorders
Keywords: Therapeutic Assessment; Psychiatry; Person-centered; Mental Health Service; Pre-therapy; Collaborative Assessment
MeSH Terms: conditions — Phobia, Social; Personality Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Naturalistic, superiority trial
Masking Description: Masking will be applied in the data analysis process
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Collaborative Assessment (MCA) (Experimental): The patients allocated to this arm will receive assessment inspired by therapeutic/collaborative assessment, as a pre-treatment to the standard psychotherapeutic treatment they will receive in the clinic.
  Interventions: Behavioral: Modified Collaborative Assessment (MCA)
- Assessment as usual (AAU) (Active Comparator): The patients allocated to this arm will receive standard assessment offered in the clinic, before proceeding to the standard psychotherapeutic treatment they will receive in the clinic.
  Interventions: Behavioral: Assessment as Usual (AAU)

INTERVENTIONS:
Behavioral: Modified Collaborative Assessment (MCA) — The Modified Collaborative Assessment (MCA) will be assessment of the patients that Is more thoroughly-done, and which will be inspired by the school of Therapeutic Assessment and Collaborative Assessment. It will include the EASE, SCID-interview, PSE, ADOS and SCIP-interviews.
  Arms: Modified Collaborative Assessment (MCA)
Behavioral: Assessment as Usual (AAU) — Assessment as usual is the standard assessment the patients will receive in the clinic. It includes one or more interviews with a mental health professional in the clinic.
  Arms: Assessment as usual (AAU)

SUMMARY:
The present study wish to compare the preliminarily effects and feasibility of Modified Collaborative Assessment (MCA) - a novel therapeutic approach to diagnostic assessment - with assessment-as-usual among patients with evasiveness as a core psychopathological feature in a randomised controlled study design.

DETAILED DESCRIPTION:
The present study wish to compare the preliminarily effects and feasibility of Modified Collaborative Assessment (MCA) - a novel therapeutic approach to diagnostic assessment - with assessment-as-usual (AAU) among patients with evasiveness as a core psychopathological feature in a randomised controlled study design.

The study will include and randomise 42 patients 1:1 to either MCA or AAU, which will be administered as a pre-treatment to the standard psychotherapeutic intervention they will receive in the psychotherapeutic clinic.

MCA will utilize standardised psychological tests administered in collaboration with the patients, in order to thorough diagnose the included patients. The tests available will be the Present State Examination (PSE), the Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD), the Screen for Cognitive Impairment in Psychiatry (SCIP), the Autism Diagnostic Observation Schedule (ADOS-2), the Examination of anomalous self-experience (EASE), the Wechsler Adult Intelligence Scale (WAIS-IV), the Level of Personality Functioning - Brief Form 2.0 (LPFS-BF), the Personality Inventory for DSM-5, 36 item version (PID-36) and the Conners´ Adult ADHD Rating Scales (CAARS).

Data are gathered through a number of questionnaires from patients prior to randomization (T0), at end of MCA (T1) and after four weeks of psychotherapy (T2) - absolute time depend on clinical logistics and timing of group therapy onset.

ELIGIBILITY:
Inclusion Criteria:

* A tentative ICD-10 diagnosis of either SAD or EPD
* Going to be offered treatment in the psychiatric community clinics in Naestved, Maribo or Slagelse

Exclusion Criteria:

* Severe physical health problems.
* Lack of spoken and written danish corresponding to 9th grade primary school.
* Eating disorder with BMI < 18
* Psychotic illness
* Active diagnosis of substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
University of Rhode Island Change Assessment Scale (URICA) | Baseline T0 (Week 1 after allocation) and T1 (end of intervention, an average of four weeks after allocation)
  The URICA is a 32-item self-report measure that includes 4 subscales measuring the motivation for change: Precontemplation, Contemplation, Action, and Maintenance. The minimum score is 32 and maximum value is 160. A higher score indicate that the patient is more ready to making changes in their life, compared to a lower.

SECONDARY OUTCOMES:
Liebowitz Social Anxiety Scale-Self- Report (LSAS) | Baseline T0 (Week 1 after allocation); T1 (end of intervention, an average of four weeks after allocation) and T2 (after one month psychotherapy)
  The 24-item LSAS-SR, includes questions pertaining to social interaction and performance situations. The LSAS-SR have shown to have good convergent, discriminant validity, and reliability. The minimum score is 48 and maximum value is 144. A higher score indicate that the patient have greater problems with anxiety, compared to a lower.

OTHER OUTCOMES:
Rosenberg Self-Esteem Scale (RSES) | Baseline T0 (Week 1 after allocation); T1 (end of intervention, an average of four weeks after allocation) and T2 (after one month psychotherapy)
  The RSES is a 10-item measure of self-esteem that includes five positive items and five negative items which are reversed scored (Rosenberg, 1965). In general, the RSES has demonstrated good convergent validity and good test-retest reliability and in similar populations of adults with social phobia, the RSES has demonstrated high internal consistency.
  The minimum score is 10 and maximum value is 40. A higher score indicate that the patient has a better self-esteem, compared to a lower.
General Self-Efficacy Scale (GSES) | Baseline T0 (Week 1 after allocation); T1 (end of intervention, an average of four weeks after allocation) and T2 (after one month psychotherapy)
  The GSE is a 10-item psychometric scale that is designed to a ssess optimistic self-beliefs to cope with a variety of difficult demands in life. In contrast to other scales that were designed to assess optimism, this one explicitly refers to personal agency, i.e., the belief that one's actions are responsible for successful outcomes.
  The minimum score is 10 and maximum value is 40. A higher score indicate that the patient feels better suited to handle difficult situations, compared to a lower.
Working Alliance Inventory (WAI) | T1 (end of intervention, an average of four weeks after allocation) and T2 (after one month psychotherapy)
  The WAI is a 12-item psychometric questionnaire that is designed to assess the therapeutic alliance between a patient and a therapist.
  The questionaire isn't scored.
Client Satisfaction Questionnaire (CSQ-8) | T1 (end of intervention, an average of four weeks after allocation) and T2 (after one month psychotherapy)
  The CSQ-8 is a self-report questionnaires constructed to measure satisfaction with services received by individuals and families.
  The minimum score is 8 and maximum value is 32. A higher score indicate that the patient is more satisfied with the treatment, compared to a lower.
National Patient Reported Outcome Measures (PROM)- Psychiatry | Baseline T0 (end of intervention, an average of four weeks after allocation); T1 (end of intervention) and T2 (after one month psychotherapy)
  The Danish National PROM is a 19-item, self-report measure covering patients own view on their mental and physical health, and level of general well-being.
  The minimum score is 19 and maximum value is 114. A higher score indicate that the patient is less burdened by his/her symptoms, compared to a lower.
Purpose-made questionary on specific feasibility-outcomes | T1 (end of intervention, an average of four weeks after allocation)
  We intend to - for the purpose of this trial - construct questionnaires evaluating the patients' and clinicians´ evaluation of the intervention.
Readiness for Psychotherapy Index | Baseline T0 (Week 1 after allocation) and T1 (end of intervention, an average of four weeks after allocation)
  The RPI is a 20-item self-report measure that uses a 5-point Likert scale to assess 7 dimensions of readiness for psychotherapy: level of distress, desire for change, willingness to work in therapy, recognition of problems as psychological, willingness to discuss personal matters, willingness to endure discomfort in therapy, and responsibility for change. The questionnaire will be translated and validated for use in a Danish mental health service population.
  The minimum score is 20 and maximum value is 100. A higher score indicate that the patient is less ready to participate in psychotherapy, compared to a lower.

CONTACTS AND LOCATIONS:
Overall Officials: Sidse Arnfred, MD PhD DMSc, Principal Investigator — Research Unit for Psychotherapy and Psychopathology, Psychiatry West, Region Zealand MHS
Locations (2):
- Denmark (2):
  - Psykiatrisk Klinik Maribo, Maribo, Region Sjælland
  - Psykiatrisk Klinik Næstved, Næstved, Region Sjælland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hovmand OR, Reinholt N, Dichmann K, Borisov R, Hjorthoj C, Arnfred S. Results of a randomized controlled superiority trial of the effect of modified collaborative assessment vs. standard assessment on patients' readiness for psychotherapy (CO-ASSM-RCT). Trials. 2024 Oct 25;25(1):716. doi: 10.1186/s13063-024-08517-8. PMID 39456051